CLINICAL TRIAL: NCT05522517
Title: A Phase 1, Single Center, Randomized, Controlled Platform Study Validating the Use of Candin as a Challenge Agent in Healthy Volunteers or Patients Given Concomitant Approved Interventions
Brief Title: A Study Validating the Use of Candin as a Challenge Agent in Healthy Participants - Intervention Specific Appendix 4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109261; 2022-001636-29 (EudraCT Number); NOPRODPANAP1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-08-18; First posted 2022-08-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Candin + Cosentyx (Experimental): Participants will receive a single dose of candin injection intradermally on Day 6 along with a single dose of saline solution injection of 0.9 percent (%) sodium chloride (NaCl) and a single dose of Cosentyx injection subcutaneously on Day 1.
  Interventions: Drug: Cosentyx; Drug: Candin
- Candin Challenge (No Intervention): All participants will receive single dose of candin injection intradermally on Day 6 along with a single dose of saline solution injection of 0.9 percent (%) sodium chloride (NaCl) administered intradermally and no Cosentyx.

INTERVENTIONS:
Drug: Cosentyx — Cosentyx injection will be administered subcutaneously.
  Other Names: Secukinumab
  Arms: Candin + Cosentyx
Drug: Candin — Candin will be administered interadermally along with NaCl solution.
  Arms: Candin + Cosentyx

SUMMARY:
The purpose of this study is to characterize the delayed-type hypersensitivity (DTH) response at the site of Candin intradermal injection in the presence of a targeted immune pathway inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilograms per meter square (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of no less than 50 kilograms (kg)
* Otherwise healthy on the basis of physical examination, medical history, and vital signs, and if required by the applicable Intervention Specific Appendix (ISA), a 12-lead electrocardiogram (ECG) performed at screening. Any abnormalities must be considered not clinically significant or consistent with the disease of interest, as specified in the applicable ISA. This determination must be recorded in the participant's source documents and initialed by the investigator
* Otherwise healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Has a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 [COVID-19]) reverse transcription polymerase chain reaction (RT-PCR) test within 72 hours prior to administration of study intervention
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 20 weeks after study intervention administration

Exclusion Criteria:

* History of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic, or mucocutaneous disturbances, unless consistent with the underlying disease of interest in the study population, if applicable
* History of any type of immunodeficiency or autoimmune disease or disease treatment associated with immune suppression or lymphopenia, unless consistent with the underlying disease of interest in the study population, if applicable. These include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenia and chronic granulomatous disease
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Known allergies, hypersensitivity, or intolerance to secukinumab or its excipients
* Has surgery planned within 20 weeks after the study intervention administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Presence and Size of Induration in Active Versus Control at the Candin Injection Site Compared to the Intra-individual Saline Control Injection Site Between 6 and 96 Hours After Candin Challenge | Day 7
  Number of participants with presence and size of induration in active versus control at the Candin injection site compared to the intra-individual saline control injection site between 6 and 96 hours after Candin challenge will be reported.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) in the Active Arm Versus the Control Arm | Up to Day 30
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs) in the Active Arm Versus the Control Arm | Up to Day 30
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.
Number of Participants with TEAEs by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) with a Frequency Threshold of 5 Percent (%) or More in the Active Arm Versus the Control Arm | Up to Day 30
  Number of participants with TEAEs by MedDRA SOC with a frequency threshold of 5% or more in the active arm versus the control arm will be reported. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency